CLINICAL TRIAL: NCT03492164
Title: Evaluating in Vivo PARP-1 Expression With 18F-FluorThanatrace Positron Emission Tomography (PET/CT) in Pancreatic Cancer
Brief Title: In Vivo PARP-1 Expression With 18F-FTT PET/CT in Pancreatic Cancer
Status: Terminated | Phase: Early Phase 1 | Type: Interventional
Why Stopped: Early analysis of images after 6 patients showed no activity of the radiotracer in this patient population.
Sponsor: Abramson Cancer Center at Penn Medicine (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: UPCC 42217
Record Dates: First submitted 2018-04-03; First posted 2018-04-10 (Actual); Last update posted 2024-06-12 (Actual); Status verified 2024-06

CONDITIONS: Pancreatic Cancer
MeSH Terms: conditions — Pancreatic Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- [18F]FluorThanatrace ([18F]FTT) (Other): 1-(4-(2-Fluoroethoxy)phenyl)-8,9-dihiydro-2,7,9a-triazabenzo[cd]azulen-6(7H)-one also known as [18F]FluorThanatrace or [18F]FTT is a positron emitting radiopharmaceutical that has been studied in animals for selective measurement of the in vivo inhibition of the PARP-1 nuclear enzyme with positron emission tomography (PET/CT).
  Interventions: Drug: [18F]FluorThanatrace ([18F]FTT)

INTERVENTIONS:
Drug: [18F]FluorThanatrace ([18F]FTT) — 1-(4-(2-Fluoroethoxy)phenyl)-8,9-dihiydro-2,7,9a-triazabenzo[cd]azulen-6(7H)-one also known as [18F]FluorThanatrace or [18F]FTT is a positron emitting radiopharmaceutical that has been studied in animals for selective measurement of the in vivo inhibition of the PARP-1 nuclear enzyme with positron emission tomography (PET/CT).
  Other Names: [18F] FTT

SUMMARY:
The investigators plan to enroll 30 evaluable patients with (1) a histological diagnosis of advanced pancreatic ductal adenocarcinoma who have demonstrated at least stable disease following ≥16 weeks of treatment with platinum-based chemotherapy and (2) who have signed consent to participate in a clinical trial that contains PARP inhibitor therapy and are anticipated to receive this treatment or (3) will receive PARP inhibitor therapy as part of their clinical care.

A pre-treatment 18F-FluorThanatrace ([18F]FTT) positron emission tomography/computed tomography (PET/CT) scan will be done prior to the start of treatment with a PARP inhibitor.

PET/CT imaging will be used to evaluate PARP-1 expression in sites of pancreatic cancer using the investigational radiotracer [18F]FTT. This is an observational study in that [18F]FTT PET/CT will not be used to direct treatment decisions. While patients and referring physicians will not be blinded to the [18F]FTT PET/CT results, treatment decisions will be made by the treating physicians based upon clinical criteria.

Patients will undergo approximately 60 minutes of dynamic scanning starting at the time of injection of [18F]FTT. This procedure will be followed by a skull base to mid-thigh scan, starting at approximately 60 minutes post injection. PET/CT imaging sessions will include an injection of approximately 10 mCi (approximate range for most studies is anticipated to be 8-12 mCi) of [18F]FTT. Data will be collected to evaluate uptake of [18F]FTT in sites of pancreatic cancer, which will be compared with PARP-1 expression in tissue, when available.

All 30 evaluable patients are expected to start PARP inhibitor therapy following the [18F]FTT PET/CT scan. It is expected that due to patient preference and time considerations, approximately 24 patients (80%) will also undergo a second (optional) scan that will be performed approximately 3 weeks (± 1 week) after therapy has started. The second scan is obtained to evaluate whether the PARP inhibitor therapy decreases [18F]FTT uptake, which would suggest PARP blocking by the therapy.

ELIGIBILITY:
Inclusion Criteria:

* Participants will be ≥ 18 years of age.
* Histologically proven pancreatic adenocarcinoma. .
* Deemed to have achieved stability following ≥16 weeks of platinum based therapy, in the opinion of an investigator
* Considered a candidate for PARP inhibitor therapy, with or without additional agents, either on a clinical trial or as part of clinical care.
* Participants must be informed of the investigational nature of this study and provide written informed consent in accordance with institutional and federal guidelines prior to study-specific procedures.

Exclusion Criteria:

* Females who are pregnant or breast feeding at the time of screening will not be eligible for this study; a urine pregnancy test will be performed in women of child-bearing potential at screening.
* Inability to tolerate imaging procedures in the opinion of an investigator or treating physician
* Serious or unstable medical or psychological conditions that, in the opinion of the investigator, would compromise the subject's safety or successful participation in the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 6 (Actual)
Dates: Start 2018-03-20 (Actual); Primary Completion 2024-06-11 (Actual); Study Completion 2024-06-11 (Actual)

PRIMARY OUTCOMES:
Number of Adverse Events | 3 years

CONTACTS AND LOCATIONS:
Overall Officials: Austin Pantel, MD, Principal Investigator — Abramson Cancer Center at Penn Medicine
Locations (1):
- Abramson Cancer Center of the University of Pennsylvania, Philadelphia, Pennsylvania, United States